CLINICAL TRIAL: NCT04937790
Title: Investigation of Effects of Core Stabilization and Computerized Wobble Board Exercise Training Programs in Patients With Heart Failure
Brief Title: Effects of Postural Balance Exercises in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Habibedurdu, Lecturer, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wobble board
Record Dates: First submitted 2021-06-02; First posted 2021-06-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Systolic Heart Failure; Diastolic Heart Failure
Keywords: wobble board; core stabilization; balance training; functionally capacity; heart failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: This study is 3 armed randomized controlled trial. Two groups will be participated exercise training, any intervention will not be applied to one group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core stabilization group (CSG) (Experimental): This arm consists core stabilization exercises including abdominal hallowing, supine bride, bride dog, side plank, curl-up and modified push up exercise. Each session is going to begin with warm-up training which consist of stretching exercise for upper-limb, lower-limb and trunk muscles, and complete with cool down exercise (same with warm-up training). Patients are going to attend one session of patient education before the first session.
  Interventions: Behavioral: Core stabilization group(CSG)
- Wobble board group ( WBG) (Experimental): This arm consists balance training exercises which performed on computerized wobble board for primarily lower limb and anti- gravity muscle. Each session is going to begin with warm-up training which consist of stretching exercise for upper-limb, lower-limb and trunk muscles, and complete with cool down exercise (same with warm-up training). Patients are going to attend one session of patient education before the first session.
  Interventions: Behavioral: Wobble board group (WBG)
- Control group (CG) (No Intervention): This arm was planned as a control group. Therefore, any intervention will not be performed. Patients in this arm going to participate only one session of patient education at the beginning of the program

INTERVENTIONS:
Behavioral: Core stabilization group(CSG) — Exercises training of this group occurs from 3 stages. In the stage 1 covering the first two weeks, core stabilization exercises are going to be applied 3 sets of 10 repetitions except side plank. Side plank is going to be performed 3 sets of 10 seconds. Stage 2 is going to include from 3 to 5 weeks. In this stage, exercises are going to be performed 3 sets of 12 repetitions except bride dog, plank and side plank. These exercises are going to be applied 3 sets of 15 seconds. Patients are going to perform exercises of stage 3 from 6 to 8 weeks. Exercises of stage 3 are going to be practiced 3 sets of 15 repetitions except bride dog, side plank and plank exercises which are going to be applied 3 set of 20 second. All stages include the same exercises except modified push-up exercise includes instead of plank exercise in stage 1. All of the exercises are going to practiced 3 days a week for 8 weeks. One of the sessions is estimated to take approximately 45-60 minutes.
  Arms: Core stabilization group (CSG)
Behavioral: Wobble board group (WBG) — Patients in this group are going to perform exercise on computerized wobble board. This device is going to provide unstable surface to patient and offer visual feedback about their movement qualities. The 8 weeks program consists of 3 stages and each stage includes six exercises. In the first stage covering the first two weeks, repetitive exercises are going to be practiced 3 sets of 10 repetitions; time controlled exercises are going to be practiced 3 sets of 20 seconds. Stage 2 is going to include from 3 to 5 weeks. In this stage, repetitive exercises are going to be performed 3 sets of 12 repetition and time controlled exercises are going to be performed 3 sets of 25 seconds. Stage 3 is going to last from 6 to 8 weeks. In this stage, repetitive exercises are going to be practiced 3 sets of 15 repetitions and time controlled exercises are going to be practiced 3 sets of 30 seconds. One of the sessions is estimated to take approximately 45-60 minutes.
  Arms: Wobble board group ( WBG)

SUMMARY:
In this study, the effects of core stabilization and computerized wobble board exercise training programs on postural balance and functional exercise capacity in patients over 60 years of age with heart failure will be investigated.

DETAILED DESCRIPTION:
This study will consist of core stabilization group (CSG), wobble board group (WBG) and control group. In CSG, exercises that focus basically on the abdominal, pelvic floor, trunk extensor and diaphragm muscles and comply with core stabilization criteria will be applied. In WBG, balance exercises which focus primarily lower limb and trunk muscles, will be performed on computerized wobble board with visual feed-back provided by computerized wobble board. In control group, no exercise will be performed, only the evaluation procedure will be applied at the beginning and 8 weeks later. It was planned to include in total of 36 patients and will be randomized them into three groups with 12 patients. Following the initial assessment, each patient will participate in a one-session patient education program. After that, patients in CSG and WBG will participate in their exercise training program which supervised by physiotherapist, 3 days a week for 8 weeks.When the exercise training programs for 8 weeks were completed, initial evaluations will be re-applied. Collected data will be analyzed with SPSS 22.0 (IBM Corp., Armonk, NY, USA) program. The differences between pre- and post-treatment evaluations will be analyzed with "paired t test" and/ or " wilcoxon test".The differences between three groups will be analyzed with one-way analysis of variance and/ or Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* Patients with heart failure who diagnosed by cardiologist
* Patients have stable drug therapy and to be clinically stable at least last three months
* Patients who signed the informed consent form

Exclusion Criteria:

* History of myocardial infarction in the last 6 months
* Acute coronary syndrome
* Un-controlled diabetes and/ or hypertension
* Severe valvular heart disease and/ or arrhythmia
* Having a pacemaker
* Severe cognitive disorder
* Severe orthopedic and/ or neurological problem
* Visual or auditory impairment
* Walking with device

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Functional balance assessment | 8 weeks
  Functional balance is going to evaluate with "berg balance scale". The scale consists of 14 items including sitting, standing up and standing up on one foot positions.Each item is scored between "0(unable)" to "4(independent) " according to success of participant. Total score is obtained by summing the scores of all items. Maximum score is 56. Scores of 0 to 20 represent balance impairment, 21 to 40 represent acceptable balance, and 41 to 56 represent good balance
Postural swing assessment | 8 weeks
  Postural swing will have been assessed using with computerized wobble board. The participant's swings on the device are measured in the antreroposterior and mediolateral directions. Measurements are performed by the device including accelerometer which has 10 degrees of tilt angle.
Functional exercise capacity assessment | 8 weeks
  Six minute walk test( 6MWT) will be applied. The test evaluates six minute walking distance in meters accordance with ATS/ ERS statements.

SECONDARY OUTCOMES:
Core stabilization assessment | 8 weeks
  "OctoCore application" is going to be used for core stabilization assessment. The application consists of two phase. The first phase is performed with single left deadline test and bird- dog exercise test is applied in second phase. Measurement of the acceleration during tests will be performed by using smart phone which has "OctoCore application" putting on mid-line of participant's fourth lumbar vertebra.
Health-related quality of life | 8 weeks
  Minnesota Living with Heart Failure questionnaire will be utilized for evaluation. The questionnaire consists of 21 items and two sub-dimension. The sub-dimensions are as follows; physical and emotional. Each item is scored between "0 (no)" to "5 (too much)". Total score changes betwen 0 and 105. Lower point demonstrates good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe DURDU, MSc, Principal Investigator — Giresun University; Rengin DEMIR, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets to be collected, will be available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Tanriverdi A, Kahraman BO, Ozsoy I, Acar S, Senturk B, Ozpelit E, Akdeniz B, Savci S. Balance performance in patients with heart failure. Heart Lung. 2020 Sep-Oct;49(5):458-462. doi: 10.1016/j.hrtlng.2020.04.004. Epub 2020 May 18. PMID 32434700
- [Result] Piraua ALT, Cavalcante BR, de Oliveira VMA, Beltrao NB, de Amorim Batista G, Pitangui ACR, Behm D, de Araujo RC. Effect of 24-week strength training on unstable surfaces on mobility, balance, and concern about falling in older adults. Scand J Med Sci Sports. 2019 Nov;29(11):1805-1812. doi: 10.1111/sms.13510. Epub 2019 Jul 26. PMID 31273863
- [Result] Granacher U, Lacroix A, Muehlbauer T, Roettger K, Gollhofer A. Effects of core instability strength training on trunk muscle strength, spinal mobility, dynamic balance and functional mobility in older adults. Gerontology. 2013;59(2):105-13. doi: 10.1159/000343152. Epub 2012 Oct 24. PMID 23108436
- [Result] Ogaya S, Ikezoe T, Soda N, Ichihashi N. Effects of balance training using wobble boards in the elderly. J Strength Cond Res. 2011 Sep;25(9):2616-22. doi: 10.1519/JSC.0b013e31820019cf. PMID 21869636
- [Derived] Durdu H, Demir R, Zeren M, Aydin E, Gunaydin ZY, Yigit Z. The Effect of Computerized Wobble Board and Core Stabilization Exercises on Balance Performance and Exercise Capacity in Patients With Heart Failure: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Aug;105(8):1429-1438. doi: 10.1016/j.apmr.2024.04.003. Epub 2024 Apr 12. PMID 38614379